CLINICAL TRIAL: NCT04987320
Title: An Open-label, Single-dose Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Olpasiran in Chinese Subjects With Elevated Serum Lipoprotein(a)
Brief Title: A Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Olpasiran in Chinese Participants With Elevated Serum Lipoprotein(a)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20190095
Record Dates: First submitted 2021-07-26; First posted 2021-08-03 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Elevated Serum Lipoprotein(a)
Keywords: Elevated serum lipoprotein(a); Olpasiran
MeSH Terms: interventions — olpasiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Olpasiran Dose A (Experimental): Participants will be administered Olpasiran dose A as a subcutaneous injection.
  Interventions: Drug: Olpasiran
- Olpasiran Dose B (Experimental): Participants will be administered Olpasiran dose B as a subcutaneous injection.
  Interventions: Drug: Olpasiran

INTERVENTIONS:
Drug: Olpasiran — Subcutaneous injection
  Other Names: AMG 890

SUMMARY:
The main objective of this study is to evaluate the pharmacokinetics (PK) of a single dose of Olpasiran in Chinese participants with elevated serum lipoprotein(a) (Lp[a]).

ELIGIBILITY:
Inclusion Criteria:

Inclusion eligibility criteria will be evaluated in 2 parts during the screening period:

* Part 1: After written informed consent is obtained, subjects will provide a blood sample for a preliminary Lp(a) assessment to determine eligibility for Part 2 screening. Subjects with Lp(a) ≥ 70 nmol/L (or approximately ≥ 27 mg/dL) will be eligible to return to the CRU Part 2 screening. Subjects not eligible to return for Part 2 screening will be screen failed.
* Part 2: Eligible subjects will complete all remaining screening procedures and tests that establish eligibility within 40 days prior to the Day 1 visit.

Part 1:

* Must be a resident in mainland China, Hong Kong, or Taiwan, and of Chinese Ancestry.
* Male or female subjects, between 18 and 60 years of age (inclusive) at the time of Screening.
* Screening serum Lp(a) ≥ 70 nmol/L (or approximately ≥ 27 mg/dL).

Part 2:

* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [e.g., suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) as assessed by the Investigator (or designee).
* Body mass index between 18 and 32 kg/m^2 (inclusive) at the time of Screening.
* Subjects who are on statin must be on a stable dose of the same statin for at least 6 weeks prior to enrollment, and plan to remain on a stable dose (i.e., no change in medication or dosage) for the duration of the study.
* Females must be of non-reproductive potential:

  a. Postmenopausal defined as: i. Age of ≥ 55 years with no menses for at least 12 months; OR ii. Age of < 55 years with no menses for at least 12 months AND with a follicle stimulating hormone (FSH) level > 40 IU/L or according to the definition of "postmenopausal range" for the laboratory involved; OR b. History of hysterectomy; OR c. History of bilateral oophorectomy.

Exclusion Criteria:

* History or clinical evidence of peripheral neuropathy.
* Currently receiving apheresis as lipid reducing therapy.
* History or clinical evidence of bleeding diathesis or any coagulation disorder, including prothrombin time (PT), activated partial thromboplastin time (APTT), or platelet count outside of the laboratory's normal reference range at screening. Subjects with PT and/or APTT values that are outside of the laboratory's normal reference range at screening may still be eligible to proceed to enrollment if the results are judged by the investigator in consultation with the study medical monitor to not be clinically significant.
* History or clinical evidence of diabetes mellitus, including a fasting glucose ≥ 125 mg/dL (6.9 mmol/L) at Screening.
* Use of any herbal medicines, vitamins or dietary supplements known to affect lipid metabolism (e.g. sigh oils > 100mg/day, red yeast extract), within 30 days prior to dosing on Day 1 and for the duration of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2022-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Queen Mary Hospital, Hong Kong, HK, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Olpasiran Low Dose: Participants were administered a single dose of olpasiran low dose as a subcutaneous injection on Day 1.
- Olpasiran High Dose: Participants were administered a single dose of olpasiran high dose as a subcutaneous injection on Day 1.
Period: Overall Study
Arm/Group | Olpasiran Low Dose | Olpasiran High Dose
Started | 12 | 12
Completed | 12 | 11
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: included all randomized participants who received olpasiran.
Groups:
- Total: Total of all reporting groups
Arm/Group | Olpasiran Low Dose | Olpasiran High Dose | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (11.23) | 49.4 (9.23) | 45.3 (10.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 12 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of Olpasiran
Description: The serum pharmacokinetic (PK) parameters of olpasiran were calculated using standard noncompartmental methods.
Time Frame: Predose, 30 and 60 minutes, 2, 3, 6, 9, 12, 24, and 36 hours postdose on Day 1 and on study Days 3, 4, 7, 15, 29, 57, and 85
Population: PK Analysis Set: included all randomized participants who received olpasiran and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Olpasiran Low Dose | Olpasiran High Dose
Number analyzed (Participants) | 12 | 12
ng/mL | 144 (55.5) | 549 (71.5)

2. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 Extrapolated to Infinity (AUCinf) of Olpasiran
Description: The serum PK parameters of olpasiran were calculated using standard noncompartmental methods.
Time Frame: as for outcome 1
Population: PK Analysis Set: included all randomized participants who received olpasiran and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Olpasiran Low Dose | Olpasiran High Dose
Number analyzed (Participants) | 12 | 12
h*ng/mL | 2660 (24.0) | 12000 (41.2)

3. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of Olpasiran
Description: The serum PK parameters of olpasiran were calculated using standard noncompartmental methods.
Time Frame: as for outcome 1
Population: PK Analysis Set: included all randomized participants who received olpasiran and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Olpasiran Low Dose | Olpasiran High Dose
Number analyzed (Participants) | 12 | 12
h*ng/mL | 2660 (24.2) | 12000 (41.3)

4. Secondary Outcome: Time to Cmax (Tmax) of Olpasiran
Description: The serum PK parameters of olpasiran were calculated using standard noncompartmental methods.
Time Frame: as for outcome 1
Population: PK Analysis Set: included all randomized participants who received olpasiran and had evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | Olpasiran Low Dose | Olpasiran High Dose
Number analyzed (Participants) | 12 | 12
hours | 3.02 [2.85 to 9.00] | 3.11 [2.88 to 12.0]

5. Secondary Outcome: Apparent Terminal Elimination Half-life (T1/2) of Olpasiran
Description: The serum PK parameters of olpasiran were calculated using standard noncompartmental methods.
Time Frame: as for outcome 1
Population: PK Analysis Set: included all randomized participants who received olpasiran and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Olpasiran Low Dose | Olpasiran High Dose
Number analyzed (Participants) | 12 | 12
hours | 6.05 (1.59) | 6.69 (1.58)

6. Secondary Outcome: Apparent Volume of Distribution During the Terminal Elimination Phase (Vz/F) of Olpasiran
Description: The serum PK parameters of olpasiran were calculated using standard noncompartmental methods.
Time Frame: as for outcome 1
Population: PK Analysis Set: included all randomized participants who received olpasiran and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Olpasiran Low Dose | Olpasiran High Dose
Number analyzed (Participants) | 12 | 12
liters | 238 (43.5) | 176 (60.2)

7. Secondary Outcome: Apparent Total Body Clearance (CL/F) of Olpasiran
Description: The serum PK parameters of olpasiran were calculated using standard noncompartmental methods.
Time Frame: as for outcome 1
Population: PK Analysis Set: included all randomized participants who received olpasiran and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Olpasiran Low Dose | Olpasiran High Dose
Number analyzed (Participants) | 12 | 12
L/h | 28.2 (24.0) | 18.8 (41.2)

8. Secondary Outcome: Number of Participants Who Experienced Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical trial participant. A TEAE was defined as an AE that starts on or after the first dose of investigational product and up to end of study.
  Clinically significant changes in clinical laboratory tests, 12-lead electrocardiograms, and vital signs were reported as AEs.
Time Frame: Up to Day 225
Population: Safety Analysis Set: included all randomized participants who received olpasiran.
Measure: Count of Participants; unit: Participants
Arm/Group | Olpasiran Low Dose | Olpasiran High Dose
Number analyzed (Participants) | 12 | 12
Participants | 12 | 10

9. Secondary Outcome: Percentage Change From Baseline in Triglycerides
Description: Participants were fasted overnight (at least 10 hours) before collection of blood samples for lipids.
Time Frame: Baseline and Days 7, 15, 57, 155 and 225
Population: Pharmacodynamic (PD) Analysis Set: included all randomized participants who received olpasiran and had evaluable PD data.
Measure: Mean (Standard Deviation); unit: percentage change in triglycerides
Arm/Group | Olpasiran Low Dose | Olpasiran High Dose
Number analyzed (Participants) | 12 | 11
percentage change in triglycerides
  Day 7 | 21.8 (30.1) | -10.0 (39.1)
  Day 15 | 10.4 (33.2) | -12.9 (22.1)
  Day 57 | 7.55 (35.1) | -2.35 (36.3)
  Day 155 | -2.87 (32.8) | -16.2 (25.3)
  Follow-up (Day 225) | 26.6 (50.7) | -10.4 (23.7)

10. Secondary Outcome: Percentage Change From Baseline in Very Low-density Lipoprotein Cholesterol (VLDL-C)
Description: Participants were fasted overnight (at least 10 hours) before collection of blood samples for lipids.
Time Frame: Baseline and Days 7, 15, 57, 155 and 225
Population: PD Analysis Set: included all randomized participants who received olpasiran and had evaluable PD data.
Measure: Mean (Standard Deviation); unit: percentage change in VLDL-C
Arm/Group | Olpasiran Low Dose | Olpasiran High Dose
Number analyzed (Participants) | 12 | 11
percentage change in VLDL-C
  Day 7 | 23.5 (37.7) | -8.43 (40.2)
  Day 15 | 13.5 (41.8) | -8.10 (32.3)
  Day 57 | 7.94 (38.3) | 4.55 (60.4)
  Day 155 | -0.165 (43.1) | -11.9 (39.0)
  Follow-up (Day 225) | 26.7 (48.4) | -7.58 (28.1)

11. Secondary Outcome: Percentage Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C)
Description: Participants were fasted overnight (at least 10 hours) before collection of blood samples for lipids.
Time Frame: Baseline and Days 7, 15, 57, 155 and 225
Population: PD Analysis Set: included all randomized participants who received olpasiran and had evaluable PD data.
Measure: Mean (Standard Deviation); unit: percentage change in LDL-C
Arm/Group | Olpasiran Low Dose | Olpasiran High Dose
Number analyzed (Participants) | 12 | 11
percentage change in LDL-C
  Day 7 | -4.17 (13.1) | 1.22 (8.36)
  Day 15 | -0.843 (14.3) | 3.97 (11.9)
  Day 57 | 0.201 (9.64) | 2.29 (9.73)
  Day 155 | -5.91 (13.5) | -3.82 (12.6)
  Follow-up (Day 225) | 2.01 (17.7) | -5.55 (10.9)

12. Secondary Outcome: Percentage Change From Baseline in High-density Lipoprotein Cholesterol (HDL-C)
Description: Participants were fasted overnight (at least 10 hours) before collection of blood samples for lipids.
Time Frame: Baseline and Days 7, 15, 57, 155 and 225
Population: PD Analysis Set: included all randomized participants who received olpasiran and had evaluable PD data.
Measure: Mean (Standard Deviation); unit: percentage change in HDL-C
Arm/Group | Olpasiran Low Dose | Olpasiran High Dose
Number analyzed (Participants) | 12 | 11
percentage change in HDL-C
  Day 7 | 3.80 (7.28) | 7.41 (6.57)
  Day 15 | 6.65 (6.18) | 11.0 (5.97)
  Day 57 | 7.17 (10.8) | 1.29 (8.40)
  Day 155 | 21.8 (11.0) | 21.3 (9.82)
  Follow-up (Day 225) | 13.9 (5.25) | 11.3 (15.3)

13. Secondary Outcome: Percentage Change From Baseline in Total Cholesterol
Description: Participants were fasted overnight (at least 10 hours) before collection of blood samples for lipids.
Time Frame: Baseline and Days 7, 15, 57, 155 and 225
Population: PD Analysis Set: included all randomized participants who received olpasiran and had evaluable PD data.
Measure: Mean (Standard Deviation); unit: percentage change in total cholesterol
Arm/Group | Olpasiran Low Dose | Olpasiran High Dose
Number analyzed (Participants) | 12 | 11
percentage change in total cholesterol
  Day 7 | 0.923 (10.2) | 0.956 (6.78)
  Day 15 | 2.45 (9.52) | 3.70 (9.03)
  Day 57 | 2.17 (7.41) | 0.879 (7.20)
  Day 155 | 1.20 (9.71) | 0.689 (8.03)
  Follow-up (Day 225) | 6.95 (9.43) | -1.82 (8.33)

14. Secondary Outcome: Percentage Change From Baseline in Apolipoprotein A1 (ApoA1)
Description: Participants were fasted overnight (at least 10 hours) before collection of blood samples for lipids.
Time Frame: Baseline and Days 7, 15, 57, 155 and 225
Population: PD Analysis Set: included all randomized participants who received olpasiran and had evaluable PD data.
Measure: Mean (Standard Deviation); unit: percentage change in ApoA1
Arm/Group | Olpasiran Low Dose | Olpasiran High Dose
Number analyzed (Participants) | 12 | 11
percentage change in ApoA1
  Day 7 | 2.86 (9.63) | 3.75 (9.46)
  Day 15 | 8.10 (5.61) | 7.95 (8.65)
  Day 57 | 0.185 (8.20) | -0.294 (8.32)
  Day 155 | 11.4 (9.46) | 9.31 (9.47)
  Follow-up (Day 225) | 18.1 (8.27) | 11.7 (14.0)

15. Secondary Outcome: Percentage Change From Baseline in Apolipoprotein B (Apo B)
Description: Participants were fasted overnight (at least 10 hours) before collection of blood samples for lipids.
Time Frame: Baseline and Days 7, 15, 57, 155 and 225
Population: PD Analysis Set: included all randomized participants who received olpasiran and had evaluable PD data.
Measure: Mean (Standard Deviation); unit: percentage change in Apo B
Arm/Group | Olpasiran Low Dose | Olpasiran High Dose
Number analyzed (Participants) | 12 | 11
percentage change in Apo B
  Day 7 | 0.0576 (11.1) | 1.41 (7.54)
  Day 15 | 2.65 (8.99) | 1.77 (9.34)
  Day 57 | 3.66 (10.0) | 1.59 (8.49)
  Day 155 | -0.834 (12.9) | -0.958 (9.01)
  Follow-up (Day 225) | 5.64 (12.4) | -1.90 (11.5)

16. Secondary Outcome: Percentage Change From Baseline in Lipoprotein-a (Lp[a])
Description: Participants were fasted overnight (at least 10 hours) before collection of blood samples for lipids.
Time Frame: Baseline and Days 2, 4, 7, 15, 29, 57, 85, 113, 155, 183 and 225
Population: PD Analysis Set: included all randomized participants who received olpasiran and had evaluable PD data.
Measure: Mean (Standard Deviation); unit: percentage change in Lp(a)
Arm/Group | Olpasiran Low Dose | Olpasiran High Dose
Number analyzed (Participants) | 12 | 12
percentage change in Lp(a)
  Day 2 | 0.245 (8.57) | -0.295 (9.84)
  Day 4 | -4.93 (11.4) | -17.6 (12.6)
  Day 7: number analyzed (Participants) | 12 | 11
  Day 7 | -32.9 (13.2) | -49.8 (16.3)
  Day 15: number analyzed (Participants) | 12 | 11
  Day 15 | -77.3 (8.46) | -84.2 (10.7)
  Day 29: number analyzed (Participants) | 12 | 11
  Day 29 | -91.0 (4.20) | -95.2 (5.50)
  Day 57: number analyzed (Participants) | 12 | 11
  Day 57 | -94.8 (3.80) | -99.2 (1.65)
  Day 85: number analyzed (Participants) | 12 | 11
  Day 85 | -91.4 (9.89) | -98.9 (1.84)
  Day 113: number analyzed (Participants) | 12 | 11
  Day 113 | -87.8 (11.1) | -97.7 (2.84)
  Day 155: number analyzed (Participants) | 12 | 11
  Day 155 | -75.8 (17.9) | -93.7 (5.13)
  Day 183: number analyzed (Participants) | 12 | 11
  Day 183 | -67.3 (18.0) | -89.1 (8.17)
  Follow-up (Day 225): number analyzed (Participants) | 12 | 11
  Follow-up (Day 225) | -55.1 (18.5) | -81.5 (11.8)

ADVERSE EVENTS:
Time Frame: Up to 225 days
Description: Safety Analysis Set: included all randomized participants who received olpasiran.
Arm/Group | Olpasiran Low Dose | Olpasiran High Dose
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12 | 1/12
Other Adverse Events (participants affected / at risk) | 11/12 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olpasiran Low Dose (N=12) | Olpasiran High Dose (N=12)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olpasiran Low Dose (N=12) | Olpasiran High Dose (N=12)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 2 (2)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 3 (3)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Dental restoration failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT04987320/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT04987320/SAP_001.pdf